CLINICAL TRIAL: NCT04859088
Title: Combining Partial Enteral Nutrition With Biologics to Optimise Induction and Maintenance Therapy for Adults With Active Ileocolonic Crohn's Disease
Brief Title: Biologics and Partial Enteral Nutrition Study
Acronym: BIOPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN21RH169
Record Dates: First submitted 2021-04-15; First posted 2021-04-26 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Crohn Disease
Keywords: Inflammatory Bowel Disease; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial Enteral Nutrition (Experimental): Patients allocated to Partial Enteral Nutrition study arm will be asked to replace 50% of their daily energy requirements with a proprietary formula (Modulen IBD, Nestle) for 6 weeks alongside standard care of treatment with adalimumab as induction therapy.
  Interventions: Dietary Supplement: Partial Enteral Nutrition
- Unrestricted diet (No Intervention): Patients allocated to unrestricted diet study arm will be asked to follow their normal diet for 6 weeks alongside standard care of treatment with adalimumab as induction therapy.

INTERVENTIONS:
Dietary Supplement: Partial Enteral Nutrition — Dietary intervention (Liquid food replacement intervention)
  Arms: Partial Enteral Nutrition

SUMMARY:
Crohn's disease (CD) is a chronic, incurable condition associated with inflammation in the gut lining. It causes diarrhoea, severe abdominal pain, poor nutrition and adversely affects the quality of life of sufferers. Two of the best treatments currently used in people with CD are drug injections and/or infusions (biologics), and a liquid-only diet using specialised milkshakes. However, treatment with biologics is only successful in approximately 40% of the patients, and although treatment with the liquid-only diet has a better safety and effectiveness profile, it is difficult for patients to stick to this as their sole source of nutrition for 6-8 weeks, particularly for adults. BIOPIC study aims to investigate whether replacing half of a habitual diet with specialised milkshakes will improve response to standard treatment with biologics in adults with CD.

DETAILED DESCRIPTION:
80 adult patients with active CD who are due to start biologic injections therapy with adalimumab as part of their standard of care for the first time will be recruited for this study. Patients will be randomly allocated to replace either half of their normal diet with nutritionally complete milkshakes or to follow their usual diet for 6 weeks. The investigators will compare the proportion of patients whose symptoms and disease markers will improve between the two groups at 6 and 12 weeks, and how many of them will remain symptoms-free for up to a year following treatment. The investigators will also explore whether the half-liquid diet will influence patients' nutrition and quality of life. Last, the investigators will investigate if gut bacteria changes and their metabolites associate with patients' eating habits and their responses to treatment with biologics.

The primary aim of the BIOPIC study is to investigate if replacement of 50% of habitual food intake with a proprietary liquid diet for 6 weeks will improve remission rates at 12 weeks in adult patients with active ileocolonic CD treated with first-line biologics (TNFα antagonists, adalimumab) as their standard treatment of care. The secondary aim is to investigate if replacement of 50% of habitual food intake with a proprietary liquid diet for 6 weeks will prolong remission in adult patients with active ileocolonic CD treated with first-line biologics (TNFα antagonists) as their standard treatment of care.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are all adults (≥16 years old) with active CD (defined as Crohn's Disease Activity Index ≥ 150) who are due to initiate standard adalimumab (TNFα antagonist) induction treatment (160 mg day 0, 80 mg at 2 weeks and then 40 mg every 2 weeks).

Exclusion Criteria:

* Inability to provide written consent to participate in the study
* Pregnant and/or breastfeeding individuals
* Presence of stoma
* Presence of short bowel syndrome
* Previous treatment with an anti-TNFα inhibitor
* Use of any other biologic therapy or oral small molecule therapy within the last 12 weeks
* Patients currently receiving oral or intravenous steroids at a dosage >20mg/day prednisolone or >9mg budesonide
* Introduction of or change in dose of immunomodulator (azathioprine, mercaptopurine, methotrexate) within the past 8 weeks
* Use of oral antibiotics within the past 4 weeks
* CD with a major fistulising or symptomatic fibrotic stricturing phenotype
* Patients tested positive for blood-borne viruses such as HIV and Hepatitis
* Patients with untreated tuberculosis (latent or active)
* Current enrolment in other studies of an investigational product or dietary intervention
* Food allergies, which do not permit participation in the study (e.g., cow's milk allergy)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index | Baseline to 52 weeks
  Comparison of Crohn's Disease Activity Index (CDAI) score (approximate range: 0-600) between the intervention (PEN) and control group (unrestricted diet).
  Higher CDAI scores indicate worse outcomes. Clinical response is defined as baseline CDAI score decrease of ≥ 70, and clinical remission is defined as CDAI score <150.

SECONDARY OUTCOMES:
Harvey-Bradshaw Index | Baseline to 52 weeks
  Comparison of Harvey-Bradshaw Index (HBI) score (approximate range: 0-50) between the intervention (PEN) and control group (unrestricted diet).
  Higher HBI scores indicate worse outcomes. Clinical response is defined as baseline HBI score decrease of ≥ 3, and clinical remission is defined as score <5]
Faecal Calprotectin | Baseline to 12 weeks
  Comparison of faecal calprotectin levels between the two groups.
  Higher scores indicate worse outcomes.
Blood C-Reactive Protein | Baseline to 12 weeks
  Comparison of blood C-reactive protein levels between the two groups.
  Abnormal values indicate worse outcomes.
Blood Erythrocyte Sedimentation Rate | Baseline to 12 weeks
  Comparison of blood erythrocyte sedimentation rates between the two groups.
  Abnormal values indicate worse outcomes.
Blood Albumin | Baseline to 12 weeks
  Comparison of blood albumin levels between the two groups.
  Abnormal values indicate worse outcomes.
Blood Haemoglobin | Baseline to 12 weeks
  Comparison of blood haemoglobin levels between the two groups.
  Abnormal values indicate worse outcomes.
Steroid-free remission | Baseline to 52 weeks
  Comparison of steroid-free remission rates between the two groups.
Dosage of biologics | Baseline to 52 weeks
  Comparison of biologics dose prescribed between the two groups.
Blood anti-drug antibodies | Baseline to 12 weeks
  Comparison of blood anti-drug antibodies between the two groups.
Blood adalimumab | Baseline to 12 weeks
  Comparison of blood levels of adalimumab (drug) between the two groups.
Micronutrient status | Baseline to 12 weeks
  Comparison of micronutrient status measured by NHS laboratories as standard care of treatment between the two groups.
  Abnormal values indicate worse outcomes.
Blood immunophenotype | Baseline to 12 weeks
  Comparison of immunophenotype profiles (characterisation of immune cells) measured with flow cytometry immunophenotyping between the two groups.
  Higher levels of specific pro-inflammatory cells indicate worse outcomes.
Self-Administered Inflammatory Bowel Disease Questionnaire | Baseline to 12 weeks
  Comparison of Self-Administered Inflammatory Bowel Disease Questionnaire (SIBDQ) scores (range: 10-70) between the two groups.
  Higher SIBDQ scores indicate better outcomes.
Body Mass Index | Baseline to 12 weeks
  Comparison of Body Mass Index (BMI) (kg/m2) between the two groups.
Body weight | Baseline to 12 weeks
  Comparison of body weight (kg) between the two groups.
Body fat mass | Baseline to 12 weeks
  Comparison of body fat mass (percent, %) measured with Bioelectrical Impedance Analysis between the two groups.
Body fat-free mass | Baseline to 12 weeks
  Comparison of body fat-free mass (percent, %) measured with Bioelectrical Impedance Analysis between the two groups.
Handgrip strength | Baseline to 12 weeks
  Comparison of handgrip strength measured with handgrip strength dynamometer between the two groups.

OTHER OUTCOMES:
Gut microbiome composition | Baseline to 12 weeks
  Comparison of gut microbiome composition measured with 16S rRNA sequencing and shotgun metagenomics between subgroups of patients.
Gut microbiome function | Baseline to 12 weeks
  Comparison of gut microbiome function measured with various targeted and untargeted bacterial metabolites (e.g. GC/LC-MS) between subgroups of patients.
3-day estimated food diary with food photography | Baseline to 6 weeks
  Comparison of prospective dietary intake measured with 3-day estimated food diaries with the assistance of food photography between subgroups of patients.
EPIC-NORFOLK Food Frequency Questionnaire | Baseline
  Comparison of retrospective dietary intake measured with 130-item EPIC-NORFOLK Food Frequency Questionnaire between subgroups of participants.
  Higher consumption/avoidance of specific food groups/products might indicate better outcomes.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Gartnavel General Hospital, Glasgow
  - The New Victoria Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked to provide written consent for their anonymised data to be made available to public repositories.